CLINICAL TRIAL: NCT05375435
Title: Efficacy and Safety of Triple Therapy Based on Prognostic Risk Stratification in Patients With Anti-MDA5 Antibody-positive Dermatomyositis: a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Efficacy and Safety of Triple Therapy in Patients With Anti-MDA5 Antibody-positive Dermatomyositis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Wenfeng Tan, Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TT-MDA5
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Dermatomyositis, Adult Type; Interstitial Lung Disease
MeSH Terms: conditions — Dermatomyositis; Lung Diseases, Interstitial | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Drug: triple therapy
- control group (Experimental)
  Interventions: Drug: dual-therapy

INTERVENTIONS:
Drug: triple therapy — high-dose glucocorticoids + cyclophosphamide + calcineurin inhibitor
  Arms: experimental group
Drug: dual-therapy — high-dose glucocorticoids + cyclophosphamide/calcineurin inhibitor
  Arms: control group

SUMMARY:
We conduct this study to investigate the efficacy of triple therapy (high-dose glucocorticoids + cyclophosphamide + calcineurin inhibitor) compared with dual-therapy regimens (high-dose glucocorticoids + cyclophosphamide/calcineurin inhibitor) and whether it reduces the risk of poor pulmonary prognosis in patients with moderate to high risk anti-MDA5+ DM.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients meet the diagnostic criteria for dermatomyositis of Bohan and Peter
* Anti-MDA5 Antibody-positive

Exclusion Criteria:

* Complicated with other connective tissue diseases
* Complicated with cardiovascular and respiratory disease caused by other reasons
* Interstitial lung disease caused by environment and drugs
* Patients with key research missing data or without informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
RPILD | 6 months
  Incidence of RP-ILD in patients after 6 months of treatment
Death | 6 months
  Mortality rate in patients after 6 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China